CLINICAL TRIAL: NCT01353482
Title: A Phase I/II Study of First Line Vorinostat With Pemetrexed-cisplatin, in Patients With Malignant Pleural Mesothelioma
Acronym: MESO-02
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: UCL CTC were informed by Merck Sharp & Dohme on 22.08.11 that support for the trial had been withdrawn in light of results from another trial with trial drug.
Sponsor: University College, London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Dean A. Fennell, Queen's University of Belfast
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCL/08/0359; 2009-013638-26 (EudraCT Number)
Record Dates: First submitted 2011-05-11; First posted 2011-05-13 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: mesothelioma; vorinostat
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Cisplatin; Pemetrexed; Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Phase II only - Arm I (Active Comparator): If the patient is randomised into the Vorinostat arm they will be given Pemetrexed (500mg/m2 iv) and Cisplatin (75mg/m2 iv) on day one of a 21 day cycle plus the dose of Vorinostat determined in the phase I study.
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Vorinostat
- Phase II only - Arm 2 (Placebo Comparator): If the patient is randomised into the placebo arm they will be given Pemetrexed (500mg/m2 iv) and Cisplatin (75mg/m2 iv) on day one of a 21 day cycle with the placebo for the same number of days as in the vorinostat arm.
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Placebo

INTERVENTIONS:
Drug: Cisplatin — Cisplatin (75mg/m2 iv) wil be administered on day one of a 21 day cycle for up to 6 cycles
Drug: Pemetrexed — Patients will be given Pemetrexed (500mg/m2 iv) on day one of a 21 day cycle for up to 6 cycles
Drug: Vorinostat — The dose and frequency of vorinostat will be determined in the Phase I study. Vorinostat will be given concurrently with Cisplatin/Pemetrexed.
  Arms: Phase II only - Arm I
Drug: Placebo — Patients randomised into the placebo arm of the trial will receive Cisplatin and Pemetrexed as standard as well as placebo.
  Arms: Phase II only - Arm 2

SUMMARY:
Mesothelioma is a relatively rare cancer which is becoming more common. It can affect one of two areas; the pleura (the lining of the lung) or the peritoneum (the lining of the abdomen). Cancer affecting the pleura is the more common of these and is called Pleural Mesothelioma. This is most commonly caused by exposure to asbestos.

Unfortunately mesothelioma is usually diagnosed at an advanced stage and so treatment is based around controlling the disease and managing the symptoms, rather than curing the disease.

The standard treatment for Advanced Malignant Pleural Mesothelioma is a combination of two anticancer drugs; Pemetrexed and Cisplatin.

The trial will look into whether there are benefits of adding a third drug called Vorinostat to the treatment.

DETAILED DESCRIPTION:
Mesothelioma is a rapidly lethal cancer which is increasing in incidence year on year. A projected doubling of cases has been predicted within the next two decades in Europe and the disease is usually diagnosed only after it has become advanced.

As yet the standard treatment for advanced mesothelioma, chemotherapy (cytotoxic drugs), is only for disease control and symptom management. A Phase I study of a drug called Vorinostat recently looked in to its effect, when given with standard cytotoxic drugs, on advanced solid tumours. The data for this study showed that this treatment caused a response in the tumours of patients with mesothelioma.

The study aims to examine the efficacy and safety of first-line vorinostat when used concurrently with cisplatin/pemetrexed.

In the proposed trial, we will initially conduct an initial run-in phase I study, to find the maximum tolerated dose, before embarking on the randomised phase II trial. The study is therefore in two stages:

Phase I study: to find the maximum tolerated dose of vorinostat in this patient group. Both safety (ie the observed number of Dose Limiting Toxicities per cohort and the overall toxicity profile) and the number of chemotherapy cycles administered will be used to determine the final dose of vorinostat to be used in the subsequent phase II study.

Randomised Phase II study: to evaluate the efficacy and safety of vorinostat (using the dose from the phase I study) versus placebo in combination with cisplatin and pemetrexed. The Phase II study will use a placebo and double-blinding to ensure that neither the patient nor the research team are aware of the allocated treatment, which should allow for accurate comparison of the two treatment arms and reduce the potential for researcher bias. Patients will be randomized 1:1 to the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of malignant pleural mesothelioma
* Measurable disease using modified RECIST criteria with at least one lesion ≥ 1cm using spiral CT in a single dimension. This scan must be within 28 days of randomisation.
* Performance status ECOG 01
* Age > 18
* Able to swallow oral medication
* Adequate haematological status
* Adequate organ function
* Negative serum or urine pregnancy test. Male subject agrees to use an acceptable method of birth control for the duration of the study and contraception must be used by women of child bearing potential.
* Ability to understand and willing to sign the written informed consent to participate (including donation of diagnostic biopsy tissue for research).
* Ability to comply with the requirements of the protocol

Exclusion Criteria:

* Other investigational or commercial agents or therapies administered with the intent of treating the patient's malignancy.
* Evidence of CNS metastases that in the opinion of the investigator should receive local treatment prior to systemic cytotoxic chemotherapy
* Uncontrolled intercurrent illness
* The patient has a history of prior malignant tumour, unless the patient has been without evidence of disease for at least three years, or the tumour was a nonmelanoma skin tumour or insitu cervix carcinoma.
* Prior exposure to vorinostat or another HDAC inhibitor is not allowed. Prior valproic acid is acceptable but only if there has been at least 30 days washout period
* Preplanned surgery or procedures that would interfere with the conduct of the study.
* Patients who have had surgery within 28 days of randomisation
* Receipt of extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks before enrolment is not allowed. However, drain site radiotherapy is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Phase I only - Dose-limiting toxicities | After 2 cycles of chemotherapy. (6 weeks after start of treatment)
Phase I only - Number of cycles of pemetrexed-cisplatin given | After 2 cycles of chemotherapy (6 weeks after start of treatment).
Phase II only - Progression free survival | At progression or patient death.
  Calculated as the time between the date of randomisation and date of first progression or death (from any cause), whichever occurs first. Patients who have not died or progressed will be censored at the date last seen alive (ie. the last assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fennell, Principal Investigator — Queen's University of Belfast

REFERENCES:
- See also: Cancer Research UK and UCL Cancer Trials Centre (Coordinating Centre) — http://www.ctc.ucl.ac.uk